CLINICAL TRIAL: NCT06490263
Title: A Phase I Clinical Trial in Healthy and Overweight/Obese Subjects to Investigate the Safety, Tolerability and Pharmacokinetics of Mulberry Twig Alkaloids
Brief Title: the Safety, Tolerability and Pharmacokinetics of Mulberry Twig Alkaloids in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Wehand-Bio Pharmaceutical Co., Ltd (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WH006-I-101
Record Dates: First submitted 2024-06-18; First posted 2024-07-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-06

CONDITIONS: Overweight and Obesity; Healthy
Keywords: Obesity Management; Hypoglycemic Agents
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- chewing or swallowing with single dose of WH006 in healthy subjects(Part One) (Experimental): Administered by chewing with meals or swallowing after meals, with a dosage of 126 milligrams, given as a single dose only in healthy subjects.
  Interventions: Drug: Experimental: Mulberry Twig Alkaloids Tablets 126 mg single dose in healthy subjects
- single dose ascending of WH006 in healthy subjects (Part Two) (Experimental): Administered by swallowing after meals with a single dose, four dose groups were performed sequentially in healthy subjects.
  Interventions: Drug: Mulberry Twig Alkaloids Tablets with single dose in healthy subjects
- multiple dose ascending of WH006 in healthy subjects (Part Three) (Experimental): Administered by swallowing after meals, taken three times daily; two dose groups were performed sequentially in healthy subjects.
  Interventions: Drug: Mulberry Twig Alkaloids Tablets with multiple dose in healthy subjects
- multiple dose ascending of WH006 in overweight or obese subjects(Part Three) (Experimental): Administered by swallowing after meals, taken three times daily; two dose groups were performed sequentially in overweight or obese subjects.
  Interventions: Drug: Mulberry Twig Alkaloids Tablets with multiple dose in overweight or obese subjects

INTERVENTIONS:
Drug: Experimental: Mulberry Twig Alkaloids Tablets 126 mg single dose in healthy subjects — Part One: Administered by chewing with meals or swallowing after meals, with a dosage of 126 milligrams, given as a single dose only.
  Other Names: WH006
  Arms: chewing or swallowing with single dose of WH006 in healthy subjects(Part One)
Drug: Mulberry Twig Alkaloids Tablets with single dose in healthy subjects — Parts Two: Administered by swallowing after meals with four distinct dosage groups.
  Other Names: WH006
  Arms: single dose ascending of WH006 in healthy subjects (Part Two)
Drug: Mulberry Twig Alkaloids Tablets with multiple dose in healthy subjects — Part Three: Administered by swallowing after meals with two distinct dosage groups, taken three times daily.
  Other Names: WH006
  Arms: multiple dose ascending of WH006 in healthy subjects (Part Three)
Drug: Mulberry Twig Alkaloids Tablets with multiple dose in overweight or obese subjects — Part Three: Administered by swallowing after meals with two distinct dosage groups, taken three times daily.
  Other Names: WH006
  Arms: multiple dose ascending of WH006 in overweight or obese subjects(Part Three)

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate safety, tolerability, and pharmacokinetics of the Mulberry Twig Alkaloids tablets (WH006) in healthy ，overweight and obesity subjects.

DETAILED DESCRIPTION:
This is a Phase I clinical trial of safety, tolerability and pharmacokinetics of the Mulberry Twig Alkaloids tablets (WH006) in healthy and overweight or obesity subjects. This trial is divided into three parts:

The first part study aims to compare the pharmacokinetics characteristics of WH006 chewing with the first bite of a standardized meal or swallowing after a standardized meal in healthy subjects.

The second part study aims to investigate the safety, tolerability and pharmacokinetics of single ascending doses of WH006 in healthy subjects.

The third part study aims to investigate the safety, tolerability and pharmacokinetics of multiple ascending doses of WH006 in both healthy participants and overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent.
2. Healthy volunteers,Body mass index between 18.5 and 24 kilogram per meter square (kg/m/m²) 18.5 inclusive). For obese or overweight participants, BMI must be at least 24 kg/m², with a requirement for some participants to have a BMI of 28 kg/m² or higher.
3. Subjects should have no history or current evidence of heart, liver, kidney, gastrointestinal, neurological, respiratory, psychiatric disorders, or metabolic abnormalities that the investigator deems requiring treatment. Vital signs, physical examination, laboratory tests, electrocardiogram (ECG), chest X-ray, abdominal ultrasound results should either be normal or show abnormalities that are deemed clinically insignificant by the attending physician.
4. Participants must not plan to become pregnant for six months following the last dose of the study drug, agree to use effective contraception to prevent pregnancy or causing pregnancy in their partner, and have no intention to donate sperm or eggs during the study period.
5. Individuals must comprehend the procedures and methods of this clinical trial, voluntarily participate and personally sign the informed consent form, demonstrating willingness to adhere to the protocol requirements and cooperate in providing biological samples according to the scheduled plan for testing.

Exclusion Criteria:

1. Secondary obesity, including conditions such as Cushing's syndrome, hypogonadism, growth hormone deficiency, hypothalamic disorders, pseudohypoparathyroidism, insulinoma, and hypothyroidism;
2. Presence of diseases exacerbating gastrointestinal bloating (e.g., Roemheld syndrome, severe hernias, intestinal obstruction, and peptic ulcers) or chronic gastrointestinal dysfunction with evident digestion and absorption disorders;
3. Diagnosis of diabetes mellitus according to the diagnostic guidelines set forth by the World Health Organization (WHO);
4. History of atopic allergic diseases or known allergies to the investigational product, its excipients, or similar medications;
5. History of orthostatic hypotension, syncope, transient loss of vision, or severe episodes of hypoglycemia;
6. Positive test results for Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (anti-HCV), Human Immunodeficiency Virus antibody (anti-HIV), or Treponema pallidum antibody (TP-Ab).
7. Participants with a history of drug abuse within 12 months prior to screening or those with positive urine tests for prohibited drugs;
8. Individuals with a history of alcohol abuse or frequent consumption (more than 14 units of alcohol per week, with 1 unit approximately equivalent to 360ml of beer, 45ml of 40% alcohol content spirits, or 150ml of wine) within 6 months prior to screening, or those with a positive breathalyzer test at screening/baseline, or unwillingness to abstain from alcohol during the study;
9. Those who smoked an average of more than 5 cigarettes per day within 3 months prior to screening, or unwilling to quit smoking during the study;
10. Individuals who donated blood (including apheresis) or experienced significant blood loss exceeding 400ml within 3 months prior to screening, received a blood transfusion or used blood products;
11. Participants who have taken part in any clinical trial within 3 months prior to screening, or plan to participate in another trial during or within 1 month after this study;
12. Individuals with a clinically significant surgical history as judged by the investigator within the screening period, or planning elective surgery between the dosing period and up to 1 month post-dosing;
13. Those who used any prescription drugs, traditional Chinese medicine, or herbal remedies within 4 weeks prior to dosing, or within 5 half-lives of any prescribed medication (whichever is longer), and/or consumed over-the-counter drugs, health supplements (excluding routine vitamin supplementation) within 2 weeks prior to dosing; those vaccinated within 4 weeks before dosing;
14. Participants who consumed excessive amounts of tea, coffee, or caffeine-containing beverages (≥8 cups, where 1 cup = 250ml) within 2 weeks prior to dosing, or who refuse to abstain from grapefruit juice or any food and drink containing alcohol and xanthines (including chocolate, tea, coffee, cola, etc.) for 48 hours before dosing and throughout the study;
15. Individuals who have been on a diet or undergone weight loss treatments within a month prior to dosing, or have made significant changes to their lifestyle habits (diet, exercise, etc.);
16. Pregnant or breastfeeding women, or those of childbearing potential who had unprotected sexual intercourse within 30 days prior to screening;
17. Participants with difficult venous access, poor peripheral venous condition, or unable to tolerate multiple blood draws, or have any contraindications to blood sampling;
18. Unwillingness or inability to follow lifestyle guidance as described in the study protocol;
19. Participants who are directly involved in this trial or are relatives (spouse, parents/legal guardians, siblings, or children) of personnel from the research center or the sponsor;
20. As judged by the investigator, individuals with conditions that may affect drug absorption, distribution, metabolism, excretion, or safety assessment, or that may reduce compliance, or those whom the investigator deems to pose a safety risk by participating in the study, as well as any other circumstances rendering them unsuitable for this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
All reported adverse events, serious adverse events and the percentage of drug-related adverse events, serious adverse events(Part Two and Part Three) | Part Two: From Day 1 to Day 4; Part Three: From Day 1 to Day 12.
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported.
To compare the Cmax of chewing or swallowing of WH006 with single dose(Part One) | Part One: From Day 1 to Day 2, Day 5 to Day 6;
  To measure the peak drug concentration of Mulberry Twig Alkaloids（1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA））with the first bite of a standardized meal or swallowing after a standardized meal
To compare the AUC0-32h of chewing or swallowing of WH006 with single dose(Part One) | Part One: From Day 1 to Day 2, Day 5 to Day 6;
  To measure the area under the concentration-time curve from time zero to time 32 hours of Mulberry Twig Alkaloids（1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA））with the first bite of a standardized meal or swallowing after a standardized meal
To compare the AUC0-inf of chewing or swallowing of WH006 with single dose(Part One) | Part One: From Day 1 to Day 2, Day 5 to Day 6;
  To measure the area under the concentration time curve from time zero to time infinity of Mulberry Twig Alkaloids（1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA））with the first bite of a standardized meal or swallowing after a standardized meal

SECONDARY OUTCOMES:
To determine the Cmax of WH006 with escalating single dose in healthy subjects(Part Two and Part Three) | Part Two: From Day 1 to Day 2;Part Three: From Day 1 to Day 2, Day 8 to Day 10.
  To measure the peak drug concentration of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating single dose in healthy subjects.
To determine the AUC0-48 of WH006 with escalating single dose in healthy subjects(Part Two and Part Three) | Part Two: From Day 1 to Day 2;Part Three: From Day 1 to Day 2, Day 8 to Day 10.
  To measure the area under the concentration-time curve from time zero to time 48 hours of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating single dose in healthy subjects.
To determine the AUC0-inf of WH006 with escalating single dose in healthy subjects(Part Two and Part Three) | Part Two: From Day 1 to Day 2;Part Three: From Day 1 to Day 2, Day 8 to Day 10.
  To measure the area under the concentration-time curve from time zero to time infinity of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating single dose in healthy subjects.
To determine the Cmax,ss of WH006 with escalating multiple dose in healthy and overweight or obese subjects(Part Three) | Part Three: From Day 1 to Day 10;
  To measure the maximum concentration at steady state of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating multiple dose in healthy and overweight or obese subjects.
To determine the Cmin,ss of WH006 with escalating multiple dose in healthy and overweight or obese subjects(Part Three) | Part Three: From Day 1 to Day 10;
  To measure the trough plasma concentration at steady state of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating multiple dose in healthy and overweight or obese subjects.
To determine the Cav,ss of WH006 with escalating multiple dose in healthy and overweight or obese subjects(Part Three) | Part Three: From Day 1 to Day 10;
  To measure the average concentration at steady state of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating multiple dose in healthy and overweight or obese subjects.
To determine the AUC0-tau of WH006 with escalating multiple dose in healthy and overweight or obese subjects(Part Three) | Part Three: From Day 1 to Day 10;
  To measure the area under the concentration-time curve from time zero to 5 hours, 14 hours and 24hours of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating multiple dose in healthy and overweight or obese subjects.
To determine the Rac of WH006 with escalating multiple dose in healthy and overweight or obese subjects(Part Three) | Part Three: From Day 1 to Day 10;
  To calculate the Rac (Cmax), Rac (AUC0-5),the Rac (AUC0-14), the Rac (AUC0-24), the Rac (AUC0-inf) with the ratio of D8 parameters and D1 parameters of Mulberry Twig Alkaloids(1-deoxynojirimycin（DNJ）, 1,4-dideoxy-1,4-imino-D-arabinitol（DAB）, Fagomine （FA）) with escalating multiple dose in healthy and overweight or obese subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Peking University First Hospital; Xia Zhao, Master, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No